CLINICAL TRIAL: NCT05822284
Title: The Role of Dynamic Circulating Tumor DNA-Molecular Residual Disease (ctDNA-MRD) Testing in Stage IIIB-C Oncogene-negative NSCLC Patients Treated With Induction Chemoimmunotherapy in the Multidisciplinary Team (MDT) Model of Diagnosis and Treatment
Brief Title: ctDNA-MRD in Stage IIIB-C NSCLC Patients Treated With Induction Chemoimmunotherapy
Status: Not yet recruiting | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Collaborators: Geneplus-Beijing Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Liu Wenliang, Professor, Second Xiangya Hospital of Central South University
Other Study IDs: LYF2023026
Record Dates: First submitted 2023-04-04; First posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with stage IIIB-C driver-negative NSCLC receiving induction chemoimmunotherapy
  Interventions: Diagnostic Test: NGS and ctDNA-MRD detection

INTERVENTIONS:
Diagnostic Test: NGS and ctDNA-MRD detection — NGS and ctDNA-MRD detection

SUMMARY:
The goal of this observational study is to explore whether ctDNA-MRD dynamic monitoring can more effectively predict the therapeutic effect of induction chemoimmunotherapy followed by surgery or non-surgical treatment for stage IIIB-C driver-negative NSCLC in the MDT model, so as to accurately guide clinical diagnosis and treatment.

DETAILED DESCRIPTION:
This study is a single-center, observational, non-interventional, prospective study. 50 patients diagnosed with stage IIIB-C driver-negative NSCLC receiving induction chemoimmunotherapy will be planned to be enrolled in the study. Pre-treatment biopsy tissues of enrolled patients will be collected for next-generation sequencing (NGS) of institutionally-developed 1021-gene panel, and personalized detection panel will be customized based on NGS testing results. Patients will be received induction chemoimmunotherapy followed by surgery or non-surgical treatment in the MDT model and ctDNA-MRD testing will be performed at prespecified time points. For patients who received surgery following induction therapy, peripheral blood will be collected in baseline, 1 day before the third cycle of neoadjuvant therapy, 1 day before surgery, 3 days after surgery and landmark time and pulmonary venous blood will be collected intraoperatively. For patients who received non-surgical treatment following induction therapy, peripheral blood will be collected in baseline, 1 day before the third cycle of neoadjuvant therapy, 1 day before non-surgical therapy and landmark time. All included patients will be regularly followed up for at least 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histopathology or cytology confirmed the non-small cell lung cancer
* Age ranging from 18 to 75
* Agree to participate in this study and sign an informed consent form
* Treatment-naive tumor
* Driver gene negativity
* According to the American Joint Committee on Cancer (AJCC) eighth edition of the Lung Cancer Staging Manual, the clinical stage is stage IIIB-C potentially resectable tumor
* The Eastern Cooperative Oncology Group (ECOG) performance status (PS) score is 0-1

Exclusion Criteria:

* Patients who cannot understand the content of the experiment and cannot cooperate, and those who refuse to sign the informed consent form
* Small cell lung cancer
* Driver gene positivity
* Tumor directly invades esophagus, heart, aorta, diaphragm, trachea, or carina, or is considered unresectable even following induction therapy
* Patients with solid organ or blood system transplantation
* Previous use of recombinant cytotoxic T-lymphocyte associated antigen 4 (CTLA-4), programmed cell death 1 (PD-1), or programmed cell death ligand 1 (PD-L1) immune checkpoint inhibitors
* Patients with interstitial lung disease
* Patients with acute or chronic infectious disease
* Pregnant and lactating women
* Patients who have undergone other clinical drug trials

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potentially resectable stage IIIB-C driver-negative NSCLC patients receiving induction chemoimmunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Predicting Progression Free Survival | up to 5 years
  Ability of dynamic ctDNA-MRD assessment to predict progression-free survival (PFS) in stage IIIB-C driver-negative NSCLC patients receiving induction chemoimmunotherapy followed by surgery or non-surgical therapy
Predicting pathologic complete response | Up to 1 year
  Ability of dynamic ctDNA-MRD assessment to predict pathologic complete response (pCR) in stage IIIB-C driver-negative NSCLC patients receiving induction chemoimmunotherapy followed by surgery
Predicting Overall Survival | up to 5 years
  Ability of dynamic ctDNA-MRD assessment to predict overall survival (OS) in stage IIIB-C driver-negative NSCLC patients receiving induction chemoimmunotherapy followed by surgery or non-surgical therapy

SECONDARY OUTCOMES:
Objective response rate(ORR) | Up to 1 year
  The proportion of patients achieved complete or partial remission according to RECIST 1.1 prior to definitive surgery.
Adverse events (AEs) | Up to 5 years
  Number of patients experiencing AEs will be recorded. An AE is defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Perioperative complications rate | Up to 3 years
  Number of patients experiencing perioperative complications will be recorded.
Health-related Quality of Life | Up to 5 years
  Health-related Quality of Life will be assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire version 3.0.
Perioperative pain evaluation | Up to 3 years
  Perioperative pain evaluation assessed by a numeric rating scale (NRS). A total of 11 points from 0 to 10 are used to describe the pain intensity. 0 means no pain, the number of points increases when the pain is stronger, and 10 means the most intense pain.
Lung cancer-related Quality of Life | Up to 5 years
  Health-related Quality of Life will be assessed by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire in Lung Cancer.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Thoracic Surgery, Second Xiangya Hospital of Central South University, China, Changsha, Hunan, China